CLINICAL TRIAL: NCT00503932
Title: A Phase I/II Trial of Proton Therapy With Concurrent Capecitabine for Locally Advanced and Recurrent Rectal Cancer
Brief Title: Proton Therapy With Capecitabine for Rectal Cancer
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: No participant enrollment.
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2005-0657
Record Dates: First submitted 2007-07-17; First posted 2007-07-19 (Estimated); Last update posted 2012-03-22 (Estimated); Status verified 2012-03

CONDITIONS: Rectal Cancer
Keywords: Rectal Cancer; Capecitabine; Proton Therapy; Adenocarcinoma of the rectum; Gastrointestinal; Proton Radiotherapy
MeSH Terms: conditions — Rectal Neoplasms | interventions — Proton Therapy; Radiotherapy; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Proton Therapy + Capecitabine (Experimental): Capecitabine 825 mg/m^2 by mouth twice daily on Proton Therapy (radiation) days.
  Interventions: Procedure: Proton Therapy; Drug: Capecitabine

INTERVENTIONS:
Procedure: Proton Therapy — Radiation therapy 1 time a day, for 5 days in a row (Monday-Friday) for 6 -7 weeks (30-35 treatments in all).
  Other Names: Proton-based radiotherapy; radiotherapy; Proton-RT; RT; XRT
Drug: Capecitabine — 825 mg/m^2 by mouth (PO) twice daily on days receive radiation.
  Other Names: Xeloda

SUMMARY:
The primary objective of the Phase I portion of this study is to evaluate the safety of a combination of capecitabine and proton therapy for patients with locally advanced or recurrent rectal cancer. The maximum tolerated dose (MTD) will be determined in the Phase I portion of this trial.

The primary objective of the Phase II portion of this study is to evaluate the local control rate in patients treated with the above regimen at the MTD.

Secondary Objectives:

1. To evaluate local tumor response in patients treated with the above regimen.
2. To evaluate the relapse-free and overall survival in patients treated with the above regimen.
3. To evaluate proton dosimetry in patients receiving this treatment.
4. To evaluate quality of life in patients receiving this therapy.

DETAILED DESCRIPTION:
Proton beams can be used to deliver a high dose of radiation to the treatment area while sparing surrounding normal tissues. Capecitabine is a drug that interferes with the growth of cancer cells.

Before you can start treatment on this study, you will have what are called "screening tests." These tests will help the doctor decide if you are eligible to take part in this study. You will have a complete physical exam. Blood (about 2 tablespoons) will be drawn for routine tests. Urine will be collected for routine tests. Chest x-rays and computed tomography (CT) scans of the abdomen (stomach area) and pelvis will be done. Women who are able to have children must have a negative blood or urine pregnancy test.

If you are found to be eligible to take part in this study, you will receive radiation therapy 1 time a day, for 5 days in a row (Monday-Friday) for 6 -7 weeks (30-35 treatments in all). You will take the chemotherapy drug, capecitabine, by mouth 2 times a day, at morning and night, on each of the days that you receive radiation therapy. These pills will not be taken on Saturday or Sunday. These pills should be taken within 30 minutes of eating and with a full glass of water.

During the study, every week you will have a physical exam and blood (about 2 teaspoons) will be drawn to check for side effects from chemotherapy and radiation therapy. You will be asked about any side effects you are experiencing.

You will be evaluated by a surgeon 4-6 weeks after the completion of treatment. Those with tumors that can be surgically removed will have surgery to remove the tumor 6-8 weeks after completion of treatment, as they would for the standard of care for their disease.

You will be taken off study if the disease gets worse or intolerable side effects occur.

Two (2) weeks after completing radiation therapy, you will have a follow-up visit. At this visit, you will have a physical exam. Blood (about 2 teaspoons) will be collected for routine tests. You will be asked about any side effects you are experiencing. Six (6) weeks after completing radiation therapy, you will have a follow-up visit. At this visit, you will have a physical exam, chest x-ray, and CT scan of your abdomen and pelvis. Blood (about 2 teaspoons) and urine will be collected for routine tests. You will be asked about any side effects you are experiencing.

After finishing treatment, you will have a follow-up visit every 3 months for the first 2 years, and every 6 months after that. At each visit, you will have a physical exam. Blood (about 2 teaspoons) and urine will be collected for routine tests. You will have a chest x-ray and CT scan of the abdomen and pelvis. You will be asked about any side effects you are experiencing.

One (1) year after you finish treatment, you will also have a colonoscopy or sigmoidoscopy. You will receive a separate consent for these procedures.

After participation in the study is over, you will have follow-up evaluation as needed for standard of care.

This is an investigational study. Capecitabine is FDA approved for treating colon cancer after surgery, and for treating metastatic colorectal cancer. The use of capecitabine with proton beam therapy in this study is investigational. About 50 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. All patients must have clinical stage T4 or recurrent adenocarcinoma of the rectum. Patients will be regarded as having clinical stage T4 if there is evidence of invasion of other structures on one or more of the following: endorectal ultrasound, pelvic CT, and physical examination, including pelvic examination
2. Histology must be confirmed with review by the Department of Pathology at UT MD Anderson Cancer Center.
3. All patients must have no distant metastatic disease in the liver, peritoneum, lungs, or paraaortic lymph nodes.
4. Patients must have a performance status (Karnofsky scale) of 70% or greater, and be able to tolerate the proposed radiation and chemotherapy regimen.
5. There are no age restrictions for this protocol.
6. Patients must have WBC > 4000 cells/mm^3, platelets > 150,000/mm^3, total serum bilirubin < 2 mg/dl, BUN <30 mg/dl, creatinine < 1.5 mg/dl and creatinine clearance > 50cc/min (estimated as calculated with Cockcroft-Gault equation).
7. Patients must have signed informed consent indicating that they are aware of the investigational nature of the study, and are aware that participation is voluntary. Patients must sign a study-specific consent form, which is attached to this protocol.

Exclusion Criteria:

1. Prior radiotherapy to the pelvis.
2. Pregnant or lactating woman. Woman of childbearing potential with either a positive or no pregnancy test at baseline. Woman / men of childbearing potential not using a reliable and appropriate contraceptive method. (Postmenopausal woman must have been amenorrheic for at least 12 months to be considered of non-childbearing potential). Patients will agree to continue contraception for 30 days from the date of the last study drug administration. Sexually active males must practice contraception during the study.
3. Treatment for other carcinomas within the last five years, except cured non-melanoma skin and treated in-situ cervical cancer.
4. Patients with uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, cardiac disease NYHA class III or IV, unstable angina pectoris, unstable cardiac arrythmia or tachycardia (heart rate > 100 beats/minute), poorly controlled hypertension (systolic blood pressure > 160 mm Hg or diastolic blood pressure > 100 mm Hg) or psychiatric illness/ social situations that would limit compliance with the study requirements are excluded.
5. Other serious uncontrolled medical conditions that the investigator feels might compromise study participation.
6. Major surgery within 4 weeks of the start of study treatment, without complete recovery.
7. Prior unanticipated severe reaction to fluoropyrimidine therapy or known hypersensitivity to 5-fluorouracil or capecitabine.
8. Patients on coumadin must be changed to Lovenox at least 1 week prior to starting capecitabine. Low dose (1 mg) coumadin is allowed.
9. Aluminium hydroxide and magnesium hydroxide-containing antacids such as Maalox must be stopped during this study.
10. Patients </= 18 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-07; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | 2 weeks after completion of radiotherapy
  MTD of a fixed dose of capecitabine (825 mg/m²) and 3 escalating doses of proton radiotherapy (5400, 5940, 6300 cobalt centiGray equivalent) as measured by dose-limiting toxicities using the continual reassessment method (CRM).

CONTACTS AND LOCATIONS:
Overall Officials: Prajnan Das, MD, Principal Investigator — M.D. Anderson Cancer Center

REFERENCES:
- See also: MD Anderson Cancer Center website — http://www.mdanderson.org